CLINICAL TRIAL: NCT02365246
Title: Interventional Trial With IgE-specific Immunoadsorption in Severe Atopic Dermatitis. Interventional Trial With IgE-specific Immunoadsorption in Severe Atopic Dermatitis.
Brief Title: Treatment of AD With IgE Specific Immunoadsorption (IGEIAAD)
Acronym: IGEIAAD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B322201421152
Record Dates: First submitted 2014-08-22; First posted 2015-02-18 (Estimated); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; immunoadsorption
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- immunoadsorption group (Experimental): All patients will be treated with 10 immunoadsorptions with an IgE-specific adsorption column :
  Interventions: Device: immunoadsorptions with an IgE-specific adsorption column

INTERVENTIONS:
Device: immunoadsorptions with an IgE-specific adsorption column — immunoadsorptions

SUMMARY:
Removal of IgE through adsorption of IgE on a specially designed column after apheresis of blood has the potential to improve the severity of atopic dermatitis.

In this study the investigators will treat patients with a severe form of Atopic dermatitis not responding or having to much side effects to systemic imunosuppressive treatment with this modality.

DETAILED DESCRIPTION:
Patients will be treated with immunoadsorption on 4 consecutive days week 1 and three consecutive days week 5 and week 9.

The clinical improvement and histological and serological tests will be evaluated.

ELIGIBILITY:
Inclusion criteria

1. Adults (> 18 year) with severe atopic dermatitis (objective SCORAD > 40)
2. Who's AD is persistent and stable since more than 1 year
3. Who signed the informed consent
4. Who are not pregnant or do not plan to become pregnant, during the immunoadsorption treatment
5. Who were treated in the recent past with phototherapy or immunosuppressive therapy ( one or more : cyclosporin A, methotrexate , azathioprine , mycophenolate , systemic corticosteroids ) and where this therapy was not sufficiently helpful, had unacceptable side effects or are contraindicated

Exclusion Criteria:

1. Patients who did not give an informed consent.
2. Patients with mild or moderate AD.
3. Patients with severe AD improving with, and tolerating, standard therapy (including phototherapy, short periods of corticosteroids, the above mentioned immunosuppressive therapies ) and having no contra-indications for these therapies
4. Pregnant women and female patients willing to become pregnant during the planned period of treatment or immediately after.
5. Having contra-indications for immunoadsorption:

   * Patients with a known allergy for the material used during immunoadsorption.
   * Severe cardiovascular diseases.
   * Severe bleeding during anticoagulation .
   * Treated with ACE-inhibitors.
   * Patients younger than18 years.
6. Having a malignant disease not under remission

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
clinical improvement (The improvement of Atopic dermatitis will be evaluated with different scales including SCORAD, EASI, LIS, DLQI) | one year
  The improvement of Atopic dermatitis will be evaluated with different scales including SCORAD, EASI, LIS, DLQI

SECONDARY OUTCOMES:
histological improvement and IgE tissue levels | one year
  we will evaluate the reduction of IgE and Fc epsilon RI expression in skin and total IgE in blood
Correlation between the therapeutic response and serum markers of disease activity . | one year
  we will evaluate serum levels and biomarkers such as TARC , MDC and TSLP during the course of the treatment
Effect of the treatment on positivity of skin prick tests. | one year
  we will evaluate skin prick reaction to dilution series of a previously positive allergen before and after treatment )
Evaluation of length of improvement | one year
  we will evaluate the duration of improvement after the last immunoadsorption and investigate if there is a correlation with drop in total IgE and / or biomarkers. The/ usefulness of supplemental adsorptionsessions will be investigated if there is an indication.

OTHER OUTCOMES:
Side effects of immunoadsorption | one year
  All side effects that appear during immunoadsorption or during the observation period after the last immunoadsorption will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Anne Morren, MD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

REFERENCES:
- [Result] Kasperkiewicz M, Schmidt E, Frambach Y, Rose C, Meier M, Nitschke M, Falk TM, Reich K, Ludwig RJ, Zillikens D. Improvement of treatment-refractory atopic dermatitis by immunoadsorption: a pilot study. J Allergy Clin Immunol. 2011 Jan;127(1):267-70, 270.e1-6. doi: 10.1016/j.jaci.2010.07.042. Epub 2010 Oct 20. No abstract available. PMID 20970174